CLINICAL TRIAL: NCT05149911
Title: Effect of a Life Coaching Intervention on the Well-being and Distress of Physicians: A Randomized Clinical Trial
Brief Title: Effect of a Life Coaching Intervention on the Well-being and Distress of Physicians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Anesthesiologists' Society (Other); University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20210617-01H
Record Dates: First submitted 2021-10-29; First posted 2021-12-08 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Distress, Emotional; Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching (Experimental): Participants randomized to the coaching group will receive a 1-hour initial professional coaching session followed by five 30-minute professional coaching sessions occurring at a goal frequency of every 2 to 3 weeks within 5 months (total of 3.5 coaching hours). All coaching sessions will be conducted individually (i.e. between one coach and one participant). Participants will be able to request coaching on any topic to individualize the intervention, but the general structure of the sessions will be standardized across participants. All coaching sessions will be performed over the phone or virtual web meeting as standard in coaching practices.
  Interventions: Behavioral: Life Coaching
- Control (No Intervention): Participants randomized to the control group will receive "no intervention" but will be asked to complete the distress and wellness survey at the same time points as participants in the intervention group. Participants in the control group will receive the life coaching intervention after the statistical analysis is completed.

INTERVENTIONS:
Behavioral: Life Coaching — Sessions with a professional life coach.
  Arms: Coaching

SUMMARY:
There is a widespread epidemic of distress and burnout (i.e., extreme distress) among Canadian physicians. Burnout is costly to physicians, patients, and healthcare organizations as it compromises physicians' own health and reduces their capacity to deliver high quality, safe care to patients. Life coaching delivered by certified coaches is a personal development tool. Life coaching has been proven to help individuals maximize their strengths and skills to handle stressors, regain control over their lives, act according to their core values, and achieve their full potential, consequently reducing their vulnerability to burnout. The investigators will evaluate life coaching for physicians' well-being in the current Canadian context. Physicians from centres in Canada will be randomly assigned to life coaching (intervention) or no coaching (control) group. The coaching group will receive a 1-hour initial coaching session followed by five 30-minute coaching sessions occurring at a frequency of every 2 to 3 weeks within 5 months (total of 3.5 coaching hours). All coaching sessions will be delivered virtually by certified life coaches. The investigators will assess the impact of coaching on physician distress and quality of life before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Registered staff physician, resident, or fellow
* Currently practicing in Canada
* (For the 'Francophone minority patients' group only) Sometimes conducts thorough consultations completely in French for French-speaking patients outside Quebec

Exclusion Criteria:

* Previously received life coaching in the last 5 years
* Currently receiving psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-11-22 (Estimated); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life score at 5 months | 5 months
  Assessed using the reduced version of the World Health Organization (WHO) Quality of Life (QOL) questionnaire (WHOQOL-BREF), one of the most widely used questionnaires for assessing adult QOL, including among healthcare professionals.

SECONDARY OUTCOMES:
Change in Burnout score at 5 months | 5 months
  Measured using the Maslach Burnout Inventory. Minimum score 0, maximum score 132. A higher score is worse, i.e., more burnout.
Change in Resilience score at 5 months | 5 months
  Measured using the Connor-Davidson Resilience Sale. Minimum score 0, maximum score 100. A higher score is better, i.e., more resilience.
Change in Job Satisfaction score at 5 months | 5 months
  Measured using the Global Job Satisfaction subscale of the Physician Job Satisfaction Scale. Minimum score 12, maximum score 60. A higher score is better, i.e., more satisfied.
Change in Job Engagement score at 5 months | 5 months
  Measured using the Utrecht Work Engagement Scale. Minimum score 0, maximum score 102. A higher score is better, i.e., better engagement.
Change in Job Empowerment and Meaning score at 5 months | Baseline and 5 months
  Measured using the Empowerment at Work Scale. Minimum score is 12, maximum score is 84. A higher score is better, i.e., higher empowerment.
Absence from work due to mental or physical illness | Baseline
  Measured as the number of days reported by participants.
Absence from work due to mental or physical illness | 5 months
  Measured as the number of days reported by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Boet, MD, PhD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No